CLINICAL TRIAL: NCT05775731
Title: Changes in Markers of Inflammation and of the Pro-thrombotic State Induced by Altered Sleep in Hospital Shift and Day Workers
Brief Title: Markers of Inflammation and of the Pro-thrombotic State in Hospital Shift and Day Workers
Acronym: IPNO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Sponsor
Other Study IDs: CCM 1788
Record Dates: First submitted 2023-02-21; First posted 2023-03-20 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2023-09

CONDITIONS: Shift-Work Related Sleep Disturbance; Inflammation; Hemostatic Disorder; Sleep Disorder
Keywords: sleep; hemostasis; inflammation; shift-work
MeSH Terms: conditions — Inflammation; Hemostatic Disorders; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma for identification of inflammatory and hemostasis markers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- shift worker: - shift worker: works at least 60 nights per year Each subject will have blood taken twice (before and after the night-shift), and will answer three questionnaires [Pittsburgh Sleep Quality Index, Generalized Anxiety Disorder-7 (GAD-7) for anxiety disorder and a general health questionnaire]
  Interventions: Diagnostic Test: Tests for markers of inflammation and activated hemostasis
- daily worker: - daily worker: does not work at night (from 8 pm to 6 am) Each subject will have blood taken once, and will answer three questionnaires (Pittsburgh Sleep Quality Index, GAD-7 for anxiety disorder and a general health questionnaire)
  Interventions: Diagnostic Test: Tests for markers of inflammation and activated hemostasis

INTERVENTIONS:
Diagnostic Test: Tests for markers of inflammation and activated hemostasis — Volunteers who do not have exclusion criteria, are invited to complete the three questionnaires and to choose a date for blood drawing based on whether they are shift workers or not. Blood is immediately processed for platelet markers, and stored for inflammation and coagulation markers
  Other Names: Questionnaires; Pittsburgh Sleep Quality Index, General Anxiety Disorder-7

SUMMARY:
The goal of this observational study is to learn if acutely and/or chronically altered sleep induces inflammation and/or a pro-thrombotic state (a tendency to form clots) in hospital workers who either work in shifts or are exclusively daily workers. The main questions it aims to answer are:

* Does chronically altered sleep induce a pro-inflammatory and pro-thrombotic state, which are steps towards cardiovascular disease, knowing that is associated with poor sleep?
* Does acutely disrupted sleep, such as that observed in night shift workers, induce a pro-inflammatory and pro-thrombotic state in otherwise healthy subjects? Participants in the study are hospital workers who either work in shifts, including night shifts, or only during the day. Sleep quality is assessed by a validated questionnaire (the Pittsburgh Sleep Quality Index). Markers of inflammation and of the pro-thrombotic state are measured at baseline and, if appropriate, after the night shift. These are markers of platelet activation, D-dimer, Interleukin-6 and endothelin 1, known to contribute and/or to suggest a condition of generalized inflammation and a tendency to form clots. Relevant information on health status is also collected for each participant.

DETAILED DESCRIPTION:
Impaired sleep (quantity and quality) is associated with a number of chronic diseases, including an increased risk of cardiovascular events. Some forms of sleep impairment such as insomnia are very frequent and can be easily identified through dedicated and validated questionnaires. The pathway through which impaired sleep heightens cardiovascular risk is not known. Some limited studies suggest activation of coagulation could follow chronic sleep impairment. Atherosclerotic plaque formation is associated with the activation of coagulation, and with chronic inflammation. It would be interesting to know if chronic or acute sleep impairment, such as that experienced by night-shift hospital workers, could induce an inflammatory and pro-thrombotic state either acutely or chronically.

To test whether these hypotheses are correct, volunteer hospital workers who either work in shifts or do not will be enrolled, to test activation of inflammation and hemostasis through established markers (platelet, inflammation and coagulation activation markers). Shift workers will be analyzed before and after a night shift.

Data on anxiety and general health (chronic disorders, medications) as well as on sleep, through validated questionnaires, will be also collected.

Two groups: night-shift workers and daily workers will be compared. Comparisons will be carried out also within night-shift workers, at baseline and after a nigh shift. Finally, subjects who sleep well and who do not sleep well will be compared, independently of shift work.

The investigators believe that if it is shown that insomnia, a frequent and often not addressed sleep disturbance, is associated with a pro-inflammatory and pro-thrombotic state in otherwise healthy workers, this finding would have important consequences, first of all in designing prospective studies on the development of cardiovascular disease in altered sleep and its prevention.

ELIGIBILITY:
Inclusion Criteria:

* Hospital worker who either works in shifts including night shifts, or only during the day

Exclusion Criteria:

* Known sleep disorder diagnosed by polysomnography and/or nocturnal saturation study
* Sleep apnea-hypopnea syndrome in C-PAP (Continuous Positive Airway Pressure) treatment
* Chronic treatment with sleep-inducers
* Chronic heart failure class NYHA III and IV
* Ischemic heart disease
* Venous thromboembolism
* Chronic anticoagulant and/or anti-platelet therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospital workers who volunteer for the study
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Sleep disorder | measurement relates to previous three months
  Evaluation of altered sleep (chronic or acute) through PSQI questionnaire

SECONDARY OUTCOMES:
Activation of inflammation and/or hemostasis | through study completion, an average of 8 months
  altered markers of inflammation and hemostasis in shift workers. The markers considered are Endothelin 1, D-dimer, IL-6, complete platelet activation and microvesicle formation

CONTACTS AND LOCATIONS:
Overall Officials: Elena M Faioni, MD, Principal Investigator — Centro Cardiologico Monzino
Locations (1):
- Centro Cardiologico Monzino, Milan, Italy

IPD SHARING:
Plan to Share IPD: No